CLINICAL TRIAL: NCT05839847
Title: Investigation of Low-intensity Focused Ultrasound for Human Anxiety Management
Brief Title: LIFU for Anxiety Management
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Polytechnic Institute and State University (Other)
Responsible Party: Principal Investigator, Wynn Legon, Assistant Professor, Virginia Polytechnic Institute and State University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 23-192
Record Dates: First submitted 2023-03-28; First posted 2023-05-03 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Participants will act as their own sham - sham vs real will be conducted in separate study visits. 2 arms exist for 2 variations of the NPU task.
Who Masked: Participant
Masking Description: Participant will experience the same setup in real and sham conditions. The gel puck used to couple the ultrasound signal will either have a blocking disk, or no blocking disk to either allow or block the ultrasound signal.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes | US Export: No

ARMS (2):
- NPU (Experimental): Participant will be presented with a series of images (cues) and sounds. Three conditions will occur - a no shock (N), predictable shock (P), and unpredictable shock (U). In P, shocks will only occur with the cue. In U, shocks will happen at any time. Participants will be told which condition they are in throughout the task. Startle sounds will occur throughout. 3 Study visits will occur - identical conditions for the participant, testing 2 brain regions and 1 sham visit.
  Interventions: Device: Low-intensity focused ultrasound; Device: Low-intensity focused ultrasound - sham
- NPU-c (Experimental): Participants will be presented with a moving line. When the line reaches a certain point - an event will occur. This event will either be a painful shock or a monetary reward. Startle sounds will occur throughout. 3 study visits will occur - identical conditions for the participant, testing 2 brain regions and 1 sham visit.
  Interventions: Device: Low-intensity focused ultrasound; Device: Low-intensity focused ultrasound - sham

INTERVENTIONS:
Device: Low-intensity focused ultrasound — A noninvasive brain stimulation device using low-intensity focused ultrasound (LIFU) - ultrasound will be used to test whether noninvasive brain stimulation can reduce reactions to sensory stimuli.
Device: Low-intensity focused ultrasound - sham — A sham condition that will mimic the application of LIFU without actually administering any ultrasound to the brain.

SUMMARY:
This study is examining the effects of noninvasive brain stimulation on anxiety. Low-intensity focused ultrasound (LIFU) will be utilized to neuromodulate the brain prior to a task (NPU). Physiological recordings will be taken throughout (EEG, EMG, HR, BP, RR, GSR).

DETAILED DESCRIPTION:
This study is a research project examining the effects of noninvasive brain stimulation on anxiety. This study will help us to better understand possible treatments for patients diagnosed with anxiety disorders. Participants will undergo a functional magnetic resonance imaging (fMRI) and a computed tomography (CT) scan, to image the bone and brain tissue. Participants will receive noninvasive brain stimulation using low-intensity focused ultrasound (LIFU) sound waves, to temporarily change brain activity. Participants will undergo a threat task involving brief (100ms) shocks (1-5mA) and startle noises. Brain signals (EEG), muscle twitch (EMG), heart rate and rhythm, blood pressure, respiration rate, and skin moisture will be monitored throughout. Participants will be asked to complete behavioral questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* High or low trait anxiety

Exclusion Criteria:

* claustrophobia
* Contraindications to MRI (implants)
* Contraindications to CT (pregnancy)
* Active medical disorder with CNS effects (e.g. Alzheimers)
* History of neurologic disorder (e.g. Parkinson's, epilepsy)
* History of head injury w/ LOC for >10 min
* History of alcohol or drug dependence
* History of current cardiovascular disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2023-12-20 (Actual); Primary Completion 2025-02-26 (Actual); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Change in EMG eye startle reflex | Through study completion, an average of 2 weeks
  Attenuated amplitude of startle reflex during uncertain and predictable threat tasks with lifu compared to sham.
Change in heart rate using ECG | Through study completion, an average of 2 weeks
  Attenuation of hear rate increases due to startle tasks in lifu compared to sham condition

CONTACTS AND LOCATIONS:
Locations (1):
- Fralin Biomedical Research Institute at VTC, Roanoke, Virginia, United States

IPD SHARING:
Plan to Share IPD: No